CLINICAL TRIAL: NCT05002361
Title: Effect of Dexamethasone Shortly Before Surgery on the Intraoperative Dose of Remifentanil in Total Knee Arthroplasty Patients Operated Under General Anesthesia: A Post-hoc Sub-study Analysis of the Randomized DEX-2-TKA Trial
Brief Title: Effect of Dexamethasone Shortly Before Surgery on the Intraoperative Dose of Remifentanil
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Naestved Hospital (Other)
Collaborators: Bispebjerg Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SM1-MG-2021
Record Dates: First submitted 2021-07-13; First posted 2021-08-12 (Actual); Last update posted 2021-08-12 (Actual); Status verified 2021-08

CONDITIONS: Perioperative Pain
MeSH Terms: interventions — Dexamethasone; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment A+B (Active Comparator): 24 mg dexamethasone i.v. perioperatively
  Interventions: Drug: Dexamethasone
- Placebo (Placebo Comparator): Placebo (isotonic saline) i.v. perioperatively
  Interventions: Drug: Isotonic saline

INTERVENTIONS:
Drug: Dexamethasone — 24 mg intravenous Dexamethasone (6 ml)
  Arms: Treatment A+B
Drug: Isotonic saline — 6 ml of isotonic saline
  Arms: Placebo

SUMMARY:
This explorative post hoc analysis included patients randomized in the DEX-2-TKA trial (NCT03506789) who were operated under general anesthesia with remifentanil and propofol. Patients having general anesthesia with sevoflurane were excluded. As the two groups receiving preoperative dexamethasone were identical at the time of outcome assessment, they were merged to one and were compared with placebo.

DETAILED DESCRIPTION:
The DEX-2-TKA was a randomized, blinded, placebo-controlled, multicenter trial in participants undergoing primary TKA conducted to investigate the effects of dexamethasone on morphine consumption, levels of postoperative pain, and harm. The methodology has been described in detail in the primary publication (ref), the protocol article and in the statistical analysis plan. In short, the trial was conducted at one private and four public Danish hospitals. Patients were randomized into one of three groups receiving either: Dexamethasone + placebo, dexamethasone + dexamethasone or placebo + placebo in a 1:1:1 ratio. The first dose of trial medication (intravenous dexamethasone 24 mg or placebo) was administered immediately after onset of anesthesia. Twenty-four hours after end of surgery, the second dose (dexamethasone 24 mg or placebo) was administered.

As the two groups receiving preoperative dexamethasone were identical at the time of outcome assessment for thi post-hoc analysis, they were merged to one and were compared with placebo yielding a ratio of 2:1 between the groups recieving dexamethsone and the placebo group.

Patients received either spinal anesthesia or general anesthesia (remifentanil and propofol were preferred). Before end of surgery all patients received ondansetron iv 4 mg. For patients in general anesthesia, sufentanil (0.3 μg/kg) was administered. All participants were provided with a patient-controlled analgesia pump (morphine 1 mg/mL, bolus 2 mg, lock-out 6 minutes, no background infusion) for 24 hours postoperatively. Additional boluses of 2 mg morphine on participant request were allowed the first hour after cessation of anesthesia. All participants received a protocolled non-opioid analgesic pain alleviation regime comprised of oral paracetamol 1 g and ibuprofen 400 mg given 1 hour before and every 6 hours after surgery and the surgeon administered local infiltration analgesia intraoperatively according to a standardized regimen.

The present explorative post hoc analysis included patients randomized in the DEX-2-TKA trial who were operated under general anesthesia with remifentanil and propofol. Patients having general anesthesia with sevoflurane were excluded.

ELIGIBILITY:
Inclusion Criteria:

* Participation in DEX-2-TKA (NCT03506789)
* General anesthesia

Exclusion Criteria:

* Spinal anestehesia
* Use of sevoflurane

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2018-09-14 (Actual); Primary Completion 2020-03-11 (Actual); Study Completion 2020-06-07 (Actual)

PRIMARY OUTCOMES:
Intraoperative use of remifentanil | During surgery (from surgical incision till last suture)
  mg

SECONDARY OUTCOMES:
Intraoperative use of propofol | During surgery (from surgical incision till last suture)
  mg
Anesthesia depth | During surgery (from surgical incision till last suture)
  Measured with bispectral index (BIS) - only for patients at Næstved
Time in post-anesthesia care unit (PACU) | Time at the PACU (from arrival at the PACU untill transfer to orthopedic ward), approximated 0-4 hours
  Minutes

CONTACTS AND LOCATIONS:
Overall Officials: Kasper S Gasbjerg, MD, Principal Investigator — Naestved Hospital
Locations (5):
- Denmark (5):
  - Gildhøj Privathospital, Brøndby
  - Bispebjerg Hospital, Copenhagen
  - Sjællands Universitetshospital, Køge, Køge
  - Næstsved Sygehus, Næstved
  - Odense Universitetshospital, Odense

REFERENCES:
- [Derived] Gantzel M, Gasbjerg KS, Hagi-Pedersen D, Meyhoff CS, Olsen MH, Mathiesen O, Jakobsen JC, Lunn TH. Effect of dexamethasone on intraoperative remifentanil dose in total knee arthroplasty surgery under general anaesthesia. Acta Anaesthesiol Scand. 2022 Oct;66(9):1070-1076. doi: 10.1111/aas.14118. Epub 2022 Aug 4. PMID 35908167